CLINICAL TRIAL: NCT03513107
Title: Osteoporosis in Egypt: Screening Tools' Re-validation and a Local Guide for the Management of the Condition in Males
Brief Title: Osteoporosis Screening Tools' Re-validation in Egypt Guide for the Management of the Condition in Males
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Saeed Salah Abduljalil Soliman, Lecturer of Family Medicine, Cairo University
Other Study IDs: 200070
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Osteoporosis
Keywords: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ospeoporosis score — * Scores will be calculated as indicated in their respective studies after collecting the data pertaining to them (Crandall, 2015); (Cass & Shepherd, 2013); (Reginster, et al., 2004); (Adler, et al., 2003); (Cadarette, et al., 2000); (Weinstein & Ulery, 2000); (Black, et al., 1998); (Lydick, et al., 1998).
  * Data will be treated as dichotomous for both DXA T-scores and screening scores (i.e. Osteoporosis (Yes or NO) versus positive/negative score).

SUMMARY:
To demonstrate the predictive ability of the different screening scores (i.e. OST, ORAI, ABONE, body weight criterion, age alone or others) and their potential use in the primary care setting.

DETAILED DESCRIPTION:
* A primary care sample of records at a local radiology center will be retrospectively reviewed and those of Egyptian adults who underwent DXA scanning will be included.
* Those with prior diagnoses that can affect bone mineral density (BMD) (i.e. prior osteoporosis, Paget's disease, osteomalacia, hyperparathyroidism, or hypogonadism) or history of using certain medications (i.e. bone-protective or anticonvulsant drugs) prior to undergoing the DXA scan will be excluded.
* Scores will be calculated as indicated in their respective studies after collecting the data pertaining to them (Crandall, 2015); (Cass & Shepherd, 2013); (Reginster, et al., 2004); (Adler, et al., 2003); (Cadarette, et al., 2000); (Weinstein & Ulery, 2000); (Black, et al., 1998); (Lydick, et al., 1998).
* Data will be treated as dichotomous for both DXA T-scores and screening scores (i.e. Osteoporosis (Yes or NO) versus positive/negative score). A 2 x 2 contingency table will be constructed and the different diagnostic test statistics (i.e. Sensitivities, specificities, Receiver operating characteristic curve) will be calculated using different Cut-off points to carry out sensitivity analyses (Moreover, different DXA sites and cut-offs will be included in the analyses). SPSS version 25 software (IBM Corp., USA) will be used for the statistical operations.
* Using an expected proportion of false negatives of 10% for sensitivity (i.e. based on the previous reported sensitivities for most tools being >90% (Crandall, 2015) and the performance of OST in Egypt of 83% (El-Masry, et al., 2015)) and a 95% confidence interval's width of 10% the needed sample size was estimated to be 138 (Browner, et al., 2013, p. 81 Table 6E). Power analysis will be calculated for any deviation from this estimation. Failure to meet sample size at the outset will be dealt with by prospectively screening new records for a period of 3 months.

Depending on the result, further recommendations and plans will be provided for possible applications and future research. All Deviations from the protocol will be justified.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing dexa scan testing.

Exclusion Criteria:

* people with prior diagnoses that can affect bone mineral density (BMD) (i.e. prior osteoporosis, Paget's disease, osteomalacia, hyperparathyroidism, or hypogonadism) or history of using certain medications (i.e. bone-protective or anticonvulsant drugs) prior to undergoing the DXA scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - A primary care sample of records at a local radiology center will be retrospectively reviewed and those of Egyptian adults who underwent DXA scanning will be included
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of osteoporosis scores | 6 months
  * Scores will be calculated as indicated in their respective studies after collecting the data pertaining to them (Crandall, 2015); (Cass & Shepherd, 2013); (Reginster, et al., 2004); (Adler, et al., 2003); (Cadarette, et al., 2000); (Weinstein & Ulery, 2000); (Black, et al., 1998); (Lydick, et al., 1998).
  * Data will be treated as dichotomous for both DXA T-scores and screening scores (i.e. Osteoporosis (Yes or NO) versus positive/negative score).

CONTACTS AND LOCATIONS:
Locations (1):
- Radiology center, Giza Egypt, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] dib, M. G., Nauroy, L. & Fuleihan, G. E., 2011. THE MIDDLE EAST & AFRICA REGIONAL AUDIT: Epidemiology, costs & burden of osteoporosis in 2011. [Online] Available at: https://www.iofbonehealth.org/sites/default/files/PDFs/Audit%20Middle%20East_Africa/Middle_East_Africa_audit.pdf [Accessed 31 /01 /2018].
- [Background] Adler RA, Tran MT, Petkov VI. Performance of the Osteoporosis Self-assessment Screening Tool for osteoporosis in American men. Mayo Clin Proc. 2003 Jun;78(6):723-7. doi: 10.4065/78.6.723. PMID 12934782
- [Background] Cadarette SM, Jaglal SB, Kreiger N, McIsaac WJ, Darlington GA, Tu JV. Development and validation of the Osteoporosis Risk Assessment Instrument to facilitate selection of women for bone densitometry. CMAJ. 2000 May 2;162(9):1289-94. PMID 10813010
- [Background] Crandall CJ. Risk Assessment Tools for Osteoporosis Screening in Postmenopausal Women: A Systematic Review. Curr Osteoporos Rep. 2015 Oct;13(5):287-301. doi: 10.1007/s11914-015-0282-z. PMID 26233285
- [Background] El-Masry, S. A., Hassan, N. E. & El-Banna, R. A., 2015. A new predictive index for osteoporosis among a sample of postmenopausal Egyptian women. Research Journal of Pharmaceutical, Biological and Chemical Sciences, 6(1), pp. 975-981.